CLINICAL TRIAL: NCT04995289
Title: Prone Position During ECMO in Covid Hypoxaemic Patient :A PROCESS-compliant Case Series From the Eastern Morocco
Brief Title: Prone Position During ECMO in Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Hypoxaemic Patient
Status: Completed | Type: Observational
Sponsor: Mohammed VI University Hospital (Other)
Responsible Party: Principal Investigator, Younes Oujidi, Principal Investigator, Mohammed VI University Hospital
Other Study IDs: MohammedVIUH
Record Dates: First submitted 2021-07-28; First posted 2021-08-06 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: SARS CoV 2 Infection; Hypoxemic Respiratory Failure
Keywords: ECMO; ARDS; Prone position; COVID; compliance
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prone position on ECMO patient — blood gas analysis before and after PP

SUMMARY:
Introduction:

The main manifestation of COVID-19 pneumonia is acute respiratory distress syndrome (ARDS), which in some cases can be more severe than intubation, extracorporeal membrane venous oxygenation (VV-ECMO) to ensure hematosis. Despite support from VV-ECMO, some patients may remain hypoxemic. One possible therapeutic procedure for these patients is the application of the prone position.

Objective:

The main aim of this study was to investigate the modification of the PaO2/FiO2 ratio, the compliance of the respiratory system in VV-ECMO with refractory hypoxemia. The secondary objective was to evaluate the safety and feasibility of the inclined position for ECMO.

Methods:

the investigators reviewed the electronic records and lists of all 23 COVID-19 patients. were placed for the first time in PP with an average duration of 16 h . patient characteristics, pre-ECMO characteristics, ventilator/ECMO settings, and changes in ventilator/ECMO settings and blood gas analysis before and after PP.

DETAILED DESCRIPTION:
The main objective of the current study was to investigate the change in PaO2/FiO2 ratio, the compliance of the respiratory system in VV-ECMO patients with persistent hypoxemia. Measurements were taken before PP, 1 h after the start of the PP, at the end of the PP cycle.

The secondary objective of this study was to assess the safety and feasibility of emergency positioning for patients with severe ARDS during ECMO treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SARS COV 2 infection complicated by ARDS, and needed a VV ECMO.
* patient who presented refractory hypoxemia during VV ECMO.

Exclusion Criteria:

* patient who has received ECMO V-A or ECMO VV for reasons other than ARDS.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 23 patients admitted to the intensive care unit of different genders and ethnicities were included.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
amelioration of PaO2/FiO2 | through study completion, an average of 1 yea
  the investigators recoordeed Blood gas analysis before and after Prone position

CONTACTS AND LOCATIONS:
Locations (1):
- younes Oujidi, Berkane, Morocco

IPD SHARING:
Plan to Share IPD: No